CLINICAL TRIAL: NCT07397481
Title: Dose Prediction for Antihypertensive Medications in Cirrhotic Patients Using Simcyp Program: Applications in Clinical Practice
Brief Title: Clinical Application of Simcyp-Guided Doses of Antihypertensive Drugs in Cirrhotic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mai Tarek, assistant lecturer, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-126
Record Dates: First submitted 2026-01-20; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Liver Cirrhosis; Arterial Hypertension
Keywords: Liver Cirrhosis; Anti- Hypertensive Drugs; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension; Hypertension, Portal | interventions — Nebivolol; Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- • Group A (n = 10): Child-Pugh class A patients received nebivolol at a dose of 5 mg once daily. (Active Comparator): Nebivolol at a dose of 5 mg (Nevilob 5 mg®, Marcyrl Pharmaceutical Industries, Egypt)
  Interventions: Drug: Nebivolol 5 mg
- • Group B (n = 10): Child-Pugh class A patients received carvedilol at a dose of 12.5 mg once daily. (Active Comparator): Carvedilol at a dose of 12.5 mg (Carvipress 12.5 mg®, Global Napi Pharmaceuticals, Egypt)
  Interventions: Drug: Carvedilol 12.5 mg
- Group C (n = 10): Child-Pugh B patients received nebivolol 2.5 mg once daily (Active Comparator): Nebivolol at a dose of 2.5 mg (Nevilob 2.5 mg®, Marcyrl Pharmaceutical Industries, Egypt)
  Interventions: Drug: Nebivolol 2.5 mg
- Group D (n = 10): Child-Pugh B patients received carvedilol 6.25 mg once daily (Active Comparator): Carvedilol at a dose of 6.25 mg (Carvipress 6.25 mg®, Global Napi Pharmaceuticals, Egypt)
  Interventions: Drug: Carvedilol 6.25 mg

INTERVENTIONS:
Drug: Nebivolol 5 mg — Nebivolol is a third-generation cardio-selective β-1 adrenergic blocker with nitric oxide-mediated vasodilatory properties and it is primarily used to treat hypertension . Nebivolol reduces intrahepatic vascular resistance by enhancing nitric oxide (NO) production within the hepatic endothelium, thereby lowering portal pressure.
  Other Names: Nevilob 5mg
  Arms: • Group A (n = 10): Child-Pugh class A patients received nebivolol at a dose of 5 mg once daily.
Drug: Carvedilol 12.5 mg — Carvedilol is used to treat hypertension and it lowers blood pressure effectively through a combination of β adrenergic blockade and α-1-mediated vasodilation. Carvedilol lowers portal pressure by β1-mediated reduction of cardiac output, β2-mediated splanchnic vasoconstriction, and additional α1-adrenergic blockade, which induces intrahepatic vasodilation, thereby reducing portal hypertension.
  Other Names: Carvipress 12.5 mg
  Arms: • Group B (n = 10): Child-Pugh class A patients received carvedilol at a dose of 12.5 mg once daily.
Drug: Nebivolol 2.5 mg — Nebivolol is a third-generation cardio-selective β-1 adrenergic blocker with nitric oxide-mediated vasodilatory properties and it is primarily used to treat hypertension . Nebivolol reduces intrahepatic vascular resistance by enhancing nitric oxide (NO) production within the hepatic endothelium, thereby lowering portal pressure.
  Other Names: Nevilob 2.5mg
  Arms: Group C (n = 10): Child-Pugh B patients received nebivolol 2.5 mg once daily
Drug: Carvedilol 6.25 mg — Carvedilol is used to treat hypertension and it lowers blood pressure effectively through a combination of β adrenergic blockade and α-1-mediated vasodilation. Carvedilol lowers portal pressure by β1-mediated reduction of cardiac output, β2-mediated splanchnic vasoconstriction, and additional α1-adrenergic blockade, which induces intrahepatic vasodilation, thereby reducing portal hypertension.
  Other Names: Carvipress 6.25 mg
  Arms: Group D (n = 10): Child-Pugh B patients received carvedilol 6.25 mg once daily

SUMMARY:
This was a prospective, open-label, randomized, parallel pilot clinical study conducted over 3 months on 50 Egyptian cirrhotic patients with arterial hypertension and portal hypertension, evaluating the real-world applicability of selected PBPK-guided dosing regimens. Patients were stratified according to Child-Pugh class (CP-A or CP-B) and randomly assigned to receive either nebivolol or carvedilol at doses corresponding to the closest commercially available strengths to Simcyp®-predicted doses.

Clinical evaluation included serial blood pressure measurements, comprising systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), and heart rate (HR). Doppler ultrasonographical assessment was performed to evaluate portal and hepatic hemodynamics, including portal vein diameter, portal vein velocity, congestion index, hepatic artery resistive index, and modified vascular liver index. Routine laboratory investigations were conducted to assess efficacy and safety and included liver function tests (serum albumin, total bilirubin, alanine aminotransferase [ALT], and aspartate aminotransferase [AST]), kidney function tests (serum creatinine and blood urea nitrogen [BUN]), and fasting blood glucose. Patients were followed on a monthly basis, with systematic documentation of adverse events throughout the study period.

DETAILED DESCRIPTION:
This was a prospective, randomized, parallel, open-label pilot clinical study conducted over three months on Egyptian cirrhotic patients with arterial hypertension and portal hypertension. Adult patients aged >18 years with confirmed liver cirrhosis, concomitant arterial hypertension, and portal hypertension without a history of variceal bleeding were eligible for inclusion. Patients with renal disorders or on dialysis, pregnancy, known hypersensitivity to the study medications, active malignancy within the previous two years, or recent use of drugs interacting with antihypertensive agents were excluded. Patients were stratified according to Child-Pugh (CP) classification into CP class A and CP class B and randomly allocated into four treatment groups to receive either nebivolol or carvedilol at doses corresponding to the closest commercially available strengths to Simcyp®-predicted doses. CP class A patients were assigned to Group A (nebivolol 5 mg once daily) or Group B (carvedilol 12.5 mg once daily), while CP class B patients were assigned to Group C (nebivolol 2.5 mg once daily) or Group D (carvedilol 6.25 mg once daily). Clinical evaluation included serial blood pressure measurements, comprising systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), and heart rate (HR), which were assessed at baseline and after 2, 4, 8, and 12 weeks of treatment. Doppler ultrasonographical assessment was performed to evaluate portal and hepatic hemodynamics, including portal vein diameter, portal vein velocity, congestion index, hepatic artery resistive index, and modified vascular liver index. Routine laboratory investigations were conducted to assess efficacy and safety and included liver function tests (serum albumin, total bilirubin, alanine aminotransferase [ALT], and aspartate aminotransferase [AST]), kidney function tests (serum creatinine and blood urea nitrogen [BUN]), CBC and fasting blood glucose. Patients were followed monthly throughout the study period, with systematic documentation of adverse events. During the study, four patients from CP class A discontinued participation and were excluded from the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age of patients > 18 years.
* Diagnosed with cirrhosis
* Have cardiovascular disease(Hypertension )
* Presence of portal hypertension
* No history of variceal bleeding

Exclusion Criteria:

* Patients with kidney disorder or dialysis
* Hypersensitivity to study medications
* Active cancer history in the last 2 years
* Taking drugs that interact with antihypertensive drugs in the last two weeks
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — yes > 18 years
Enrollment: 40 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Management of arterial hypertension | 3 month
  by measuring Systolic and diastolic blood pressure (mmHg)

SECONDARY OUTCOMES:
Adverse Effects Monitoring | 3 months
  Adverse effects including headache, gastrointestinal disorders, weakness, shortness of breath, and hyperglycemia will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mai Tarek Hamed, BSc (Pharmacy), Principal Investigator — Clinical Pharmacy Department, Faculty of Pharmacy, Kafrelsheikh University; Ahmed A Ali, PhD, Study Director — Clinical Pharmacy Department, Faculty of Pharmacy, Kafrelsheikh University
Locations (1):
- Kafrelsheikh University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li T, Ke W, Sun P, Chen X, Belgaumkar A, Huang Y, Xian W, Li J, Zheng Q. Carvedilol for portal hypertension in cirrhosis: systematic review with meta-analysis. BMJ Open. 2016 May 4;6(5):e010902. doi: 10.1136/bmjopen-2015-010902. PMID 27147389
- See also: Carvedilol for portal hypertension in cirrhosis: systematic review with meta-analysis — https://pubmed.ncbi.nlm.nih.gov/27147389/